CLINICAL TRIAL: NCT02328898
Title: A Prospective, Multi-Center, Open Label, Randomized Controlled, Two Arm Study Evaluating Safety and Efficacy of the Permanent Polymer Zotarolimus Eluting Stent Resolute Integrity Compared to the Polymer Free Amphilimus Eluting Stent Cre8
Brief Title: Randomized "All-comer" Evaluation of a Permanent Polymer Resolute Integrity Stent Versus a Polymer Free Cre8 Stent
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Pieter Stella, M.D. PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-244/M
Record Dates: First submitted 2014-09-16; First posted 2014-12-31 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Stable Angina Pectoris; Acute Coronary Syndrome
Keywords: Polymer free stent; percutaneous coronary intervention
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cre8 stent (Experimental): PCI with the Polymer Free Amphilimus Eluting Stent 'Cre8™'
  Interventions: Device: Cre8 Stent
- Resolute Integrity Stent (Active Comparator): Comparison of the Cre8 stent with the Permanent Polymer Zotarolimus Eluting Stent 'Resolute Integrity™'
  Interventions: Device: Resolute Integrity stent

INTERVENTIONS:
Device: Cre8 Stent — Comparison of the Resolute Integrity stent with the Cre8 stent.
  Other Names: Resolute Integrity Stent
  Arms: Cre8 stent
Device: Resolute Integrity stent
  Arms: Resolute Integrity Stent

SUMMARY:
The study objective is to assess the safety and efficacy of the Permanent Polymer Zotarolimus-Eluting Stent Resolute Integrity™ to the Polymer Free Amphilimus-Eluting Stent Cre8™ compared in an all-comer patient population. 1 month of dual antiplatelet duration will be applied in stable angina pectoris patients. Myocardial infarction patient population will be treated with 12 months of dual antiplatelet therapy.

DETAILED DESCRIPTION:
A Prospective, Multi-Center, Open Label, Randomized Controlled, two-arm Study to Evaluate the Safety and Efficacy of the Permanent Polymer Zotarolimus Eluting Stent 'Resolute Integrity™' Compared to Polymer Free Amphilimus Eluting Stent 'Cre8'. Dual Antiplatelet Therapy duration of 1 Month will be applied in stable angina pectoris patient population. Myocardial infarction patient population will be treated with 12 months of dual antiplatelet therapy (DAPT).

One thousand five hundred thirty-two (1532) patients (1:1 randomization Cre8 stent: Resolute Integrity™ stent) will be enrolled in the study, with clinical follow-up at 12 months to assess the primary end point.

After a period of 12 months, a clinical registry will be implemented Information will be collected at 3-years post procedure.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. All-comer patients aged 18 years and older
2. Patient has been informed of the nature of the trial and agrees to its provisions and has provided either oral during emergency procedure, followed by written informed consent, or written informed consent in case of an elective procedure as approved by the Medical Research Ethics Committee (MREC) of the respective investigational site
3. Patient is eligible, according to heart team decision if applicable, for PCI with implantation of a drug-eluting stent (DES)
4. Patient has clinical evidence of ischemic heart disease, angina pectoris, myocardial infarction, or silent ischemia

Angiographic Inclusion Criteria:

1. All de-novo lesions and all restenotic lesions (whether native coronary or bypass graft), not amenable for treatment with drug eluting balloons
2. All lesions types are allowed: calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), thrombus, chronic total occlusion (CTO; randomized after successful wire crossing and pre-dilatation), bifurcation lesions, ostial lesions, bypass graft (venous and arterial) lesions and left main.
3. There is no limit for lesion length; overlapping stents are allowed, or number of lesions or diseased vessels.
4. Target vessel size reference (visual estimation) between 2.5 mm and 4.5 mm.

Exclusion Criteria:

1. Inability to provide informed consent
2. Participation in another study for intracoronary stents that had not reached its primary endpoint
3. Planned surgery within the next 3 months
4. Known intolerance to P2Y12 receptor antagonist that would prevent adherence to DAPT, or intolerance to aspirin, clopidogrel, Ticagrelor, Prasugrel, heparin/bivalirudin, contrast agent (that cannot be adequately premedicated) or component of DES
5. Female of childbearing potential, who are pregnant or are planning to become pregnant
6. Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1532 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 and 36 months
  Cardiac death, vessel-related myocardial infarction (QWMI and NQWMI), target lesion revascularization by CABG or PCI

SECONDARY OUTCOMES:
Net Adverse Clinical Events (NACE) | 12 and 36 months
  defined as composite of any death, stroke, myocardial infarction, any unplanned repeated revascularization and bleeding (BARC 3a and above)
Target lesion failure (TLF) | 12 and 36 months
  separate components of the primary endpoint; cardiac death, vessel related myocardial infarction (QWMI and NQWMI), target lesion revascularization by CABG or PCI
Target vessel revascularization by CABG or PCI (TVR) | 12 and 36 months
Stent thrombosis | 12 and 36 months
Device, lesion and procedure success at time of baseline procedure | 12 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter R Stella, M.D., PhD, Principal Investigator — UMC Utrecht, the Netherlands
Locations (3):
- Institute of Cardiac Surgery and Interventional Cardiology, Luxembourg, Luxembourg
- Netherlands (2):
  - Zuyderland Medical Centre, Heerlen
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] van Hemert ND, Stella PR, Rozemeijer R, Stein M, Frambach P, Kraaijeveld AO, Rittersma SZ, Meijs TA, Leenders GEH, van der Harst P, Agostoni P, Voskuil M; ReCre8 Study Investigators. High bleeding risk in patients undergoing percutaneous coronary intervention with drug-eluting stent implantation: ReCre8 subanalysis. Am Heart J Plus. 2022 Nov 9;24:100227. doi: 10.1016/j.ahjo.2022.100227. eCollection 2022 Dec. PMID 38560639
- [Derived] van Hemert ND, Voskuil M, Rozemeijer R, Stein M, Frambach P, Pereira B, Rittersma SZ, Kraaijeveld AO, Leenders GEH, Timmers L, van der Harst P, Agostoni P, Stella PR; ReCre8 Study Investigators. 3-Year Clinical Outcomes After Implantation of Permanent-Polymer Versus Polymer-Free Stent: ReCre8 Landmark Analysis. JACC Cardiovasc Interv. 2021 Nov 22;14(22):2477-2486. doi: 10.1016/j.jcin.2021.08.078. PMID 34794654
- [Derived] Rozemeijer R, Stein M, Voskuil M, van den Bor R, Frambach P, Pereira B, Koudstaal S, Leenders GE, Timmers L, Rittersma SZ, Kraaijeveld AO, Agostoni P, Roes KC, Doevendans PA, Stella PR; ReCre8 Study Investigators. Randomized All-Comers Evaluation of a Permanent Polymer Zotarolimus-Eluting Stent Versus a Polymer-Free Amphilimus-Eluting Stent. Circulation. 2019 Jan 2;139(1):67-77. doi: 10.1161/CIRCULATIONAHA.118.037707. PMID 30586704